CLINICAL TRIAL: NCT02054806
Title: Phase IB Study of Pembrolizumab (MK-3475) in Subjects With Select Advanced Solid Tumors
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Advanced Solid Tumors (MK-3475-028/KEYNOTE-28)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-028; 142515 (Registry Identifier: JAPIC-CTI); MK-3475-028 (Other: Merck); KEYNOTE-28 (Other: Merck); 2013-004507-39 (EudraCT Number)
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 10 mg/kg, intravenously (IV), once every 2 weeks (Q2W) for up to ~2 years
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This study will assess the efficacy and safety of pembrolizumab (MK-3475) administered to participants with incurable advanced biomarker-positive solid tumors that have not responded to current therapy or for which current therapy is not appropriate.

The study hypothesis is that administration of pembrolizumab to participants with some types of solid tumors will result in a clinically meaningful response rate.

DETAILED DESCRIPTION:
Qualified participants who complete up to ~2 years of pembrolizumab treatment but progress after discontinuation may be eligible for a second course of pembrolizumab for up to ~1 additional year, at the Investigator's discretion. Per protocol, response or progression during this second course will not count towards efficacy outcome measures and adverse events during this second course will not count towards safety outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally-advanced and/or metastatic solid malignancy that is incurable, and has failed prior standard therapy or for which standard therapy is not appropriate
* Have biomarker-positive solid tumor
* Have measurable disease based on Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
* Adequate organ function
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication
* Male participants of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study medication through 120 days after the last dose of study medication

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Prior anti-cancer therapy with a monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or not recovered from adverse events due to mAbs administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks (12 weeks for measurable sites of central nervous system [CNS] disease) prior to study Day 1 or not recovered from adverse events due to a previously administered agent
* Known additional malignancy that is progressing or requires active treatment excepting basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer
* Known active CNS metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has evidence of interstitial lung disease or a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has previously participated in any other pembrolizumab (MK-3475) trial, or received prior therapy with an anti-PD-1, anti-PD-L1, and anti-PD-L2 (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or Hepatitis C
* Has received a live vaccine within 30 days of planned start of study medication. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Alley EW, Lopez J, Santoro A, Morosky A, Saraf S, Piperdi B, van Brummelen E. Clinical safety and activity of pembrolizumab in patients with malignant pleural mesothelioma (KEYNOTE-028): preliminary results from a non-randomised, open-label, phase 1b trial. Lancet Oncol. 2017 May;18(5):623-630. doi: 10.1016/S1470-2045(17)30169-9. Epub 2017 Mar 11. PMID 28291584
- [Result] Ott PA, Piha-Paul SA, Munster P, Pishvaian MJ, van Brummelen EMJ, Cohen RB, Gomez-Roca C, Ejadi S, Stein M, Chan E, Simonelli M, Morosky A, Saraf S, Emancipator K, Koshiji M, Bennouna J. Safety and antitumor activity of the anti-PD-1 antibody pembrolizumab in patients with recurrent carcinoma of the anal canal. Ann Oncol. 2017 May 1;28(5):1036-1041. doi: 10.1093/annonc/mdx029. PMID 28453692
- [Result] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Result] Ott PA, Elez E, Hiret S, Kim DW, Morosky A, Saraf S, Piperdi B, Mehnert JM. Pembrolizumab in Patients With Extensive-Stage Small-Cell Lung Cancer: Results From the Phase Ib KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 1;35(34):3823-3829. doi: 10.1200/JCO.2017.72.5069. Epub 2017 Aug 16. PMID 28813164
- [Result] Doi T, Piha-Paul SA, Jalal SI, Saraf S, Lunceford J, Koshiji M, Bennouna J. Safety and Antitumor Activity of the Anti-Programmed Death-1 Antibody Pembrolizumab in Patients With Advanced Esophageal Carcinoma. J Clin Oncol. 2018 Jan 1;36(1):61-67. doi: 10.1200/JCO.2017.74.9846. Epub 2017 Nov 8. PMID 29116900
- [Result] Frenel JS, Le Tourneau C, O'Neil B, Ott PA, Piha-Paul SA, Gomez-Roca C, van Brummelen EMJ, Rugo HS, Thomas S, Saraf S, Rangwala R, Varga A. Safety and Efficacy of Pembrolizumab in Advanced, Programmed Death Ligand 1-Positive Cervical Cancer: Results From the Phase Ib KEYNOTE-028 Trial. J Clin Oncol. 2017 Dec 20;35(36):4035-4041. doi: 10.1200/JCO.2017.74.5471. Epub 2017 Nov 2. PMID 29095678
- [Result] O'Neil BH, Wallmark JM, Lorente D, Elez E, Raimbourg J, Gomez-Roca C, Ejadi S, Piha-Paul SA, Stein MN, Abdul Razak AR, Dotti K, Santoro A, Cohen RB, Gould M, Saraf S, Stein K, Han SW. Safety and antitumor activity of the anti-PD-1 antibody pembrolizumab in patients with advanced colorectal carcinoma. PLoS One. 2017 Dec 28;12(12):e0189848. doi: 10.1371/journal.pone.0189848. eCollection 2017. PMID 29284010
- [Result] Cohen RB, Delord JP, Doi T, Piha-Paul SA, Liu SV, Gilbert J, Algazi AP, Damian S, Hong RL, Le Tourneau C, Day D, Varga A, Elez E, Wallmark J, Saraf S, Thanigaimani P, Cheng J, Keam B. Pembrolizumab for the Treatment of Advanced Salivary Gland Carcinoma: Findings of the Phase 1b KEYNOTE-028 Study. Am J Clin Oncol. 2018 Nov;41(11):1083-1088. doi: 10.1097/COC.0000000000000429. PMID 29462123
- [Result] Rugo HS, Delord JP, Im SA, Ott PA, Piha-Paul SA, Bedard PL, Sachdev J, Le Tourneau C, van Brummelen EMJ, Varga A, Salgado R, Loi S, Saraf S, Pietrangelo D, Karantza V, Tan AR. Safety and Antitumor Activity of Pembrolizumab in Patients with Estrogen Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer. Clin Cancer Res. 2018 Jun 15;24(12):2804-2811. doi: 10.1158/1078-0432.CCR-17-3452. Epub 2018 Mar 20. PMID 29559561
- [Result] Ott PA, Bang YJ, Berton-Rigaud D, Elez E, Pishvaian MJ, Rugo HS, Puzanov I, Mehnert JM, Aung KL, Lopez J, Carrigan M, Saraf S, Chen M, Soria JC. Safety and Antitumor Activity of Pembrolizumab in Advanced Programmed Death Ligand 1-Positive Endometrial Cancer: Results From the KEYNOTE-028 Study. J Clin Oncol. 2017 Aug 1;35(22):2535-2541. doi: 10.1200/JCO.2017.72.5952. Epub 2017 May 10. PMID 28489510
- [Result] Varga A, Piha-Paul S, Ott PA, Mehnert JM, Berton-Rigaud D, Morosky A, Yang P, Ruman J, Matei D. Pembrolizumab in patients with programmed death ligand 1-positive advanced ovarian cancer: Analysis of KEYNOTE-028. Gynecol Oncol. 2019 Feb;152(2):243-250. doi: 10.1016/j.ygyno.2018.11.017. Epub 2018 Dec 3. PMID 30522700
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] Reardon DA, Kim TM, Frenel JS, Simonelli M, Lopez J, Subramaniam DS, Siu LL, Wang H, Krishnan S, Stein K, Massard C. Treatment with pembrolizumab in programmed death ligand 1-positive recurrent glioblastoma: Results from the multicohort phase 1 KEYNOTE-028 trial. Cancer. 2021 May 15;127(10):1620-1629. doi: 10.1002/cncr.33378. Epub 2021 Jan 26. PMID 33496357
- [Derived] Piha-Paul SA, Oh DY, Ueno M, Malka D, Chung HC, Nagrial A, Kelley RK, Ros W, Italiano A, Nakagawa K, Rugo HS, de Braud F, Varga AI, Hansen A, Wang H, Krishnan S, Norwood KG, Doi T. Efficacy and safety of pembrolizumab for the treatment of advanced biliary cancer: Results from the KEYNOTE-158 and KEYNOTE-028 studies. Int J Cancer. 2020 Oct 15;147(8):2190-2198. doi: 10.1002/ijc.33013. Epub 2020 May 2. PMID 32359091
- [Derived] Mehnert JM, Bergsland E, O'Neil BH, Santoro A, Schellens JHM, Cohen RB, Doi T, Ott PA, Pishvaian MJ, Puzanov I, Aung KL, Hsu C, Le Tourneau C, Hollebecque A, Elez E, Tamura K, Gould M, Yang P, Stein K, Piha-Paul SA. Pembrolizumab for the treatment of programmed death-ligand 1-positive advanced carcinoid or pancreatic neuroendocrine tumors: Results from the KEYNOTE-028 study. Cancer. 2020 Jul 1;126(13):3021-3030. doi: 10.1002/cncr.32883. Epub 2020 Apr 22. PMID 32320048
- [Derived] Mehnert JM, Varga A, Brose MS, Aggarwal RR, Lin CC, Prawira A, de Braud F, Tamura K, Doi T, Piha-Paul SA, Gilbert J, Saraf S, Thanigaimani P, Cheng JD, Keam B. Safety and antitumor activity of the anti-PD-1 antibody pembrolizumab in patients with advanced, PD-L1-positive papillary or follicular thyroid cancer. BMC Cancer. 2019 Mar 4;19(1):196. doi: 10.1186/s12885-019-5380-3. PMID 30832606
- [Derived] Ott PA, Bang YJ, Piha-Paul SA, Razak ARA, Bennouna J, Soria JC, Rugo HS, Cohen RB, O'Neil BH, Mehnert JM, Lopez J, Doi T, van Brummelen EMJ, Cristescu R, Yang P, Emancipator K, Stein K, Ayers M, Joe AK, Lunceford JK. T-Cell-Inflamed Gene-Expression Profile, Programmed Death Ligand 1 Expression, and Tumor Mutational Burden Predict Efficacy in Patients Treated With Pembrolizumab Across 20 Cancers: KEYNOTE-028. J Clin Oncol. 2019 Feb 1;37(4):318-327. doi: 10.1200/JCO.2018.78.2276. Epub 2018 Dec 13. PMID 30557521
- [Derived] Hansen AR, Massard C, Ott PA, Haas NB, Lopez JS, Ejadi S, Wallmark JM, Keam B, Delord JP, Aggarwal R, Gould M, Yang P, Keefe SM, Piha-Paul SA. Pembrolizumab for advanced prostate adenocarcinoma: findings of the KEYNOTE-028 study. Ann Oncol. 2018 Aug 1;29(8):1807-1813. doi: 10.1093/annonc/mdy232. PMID 29992241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a histologically- or cytologically-confirmed diagnosis of 20 advanced (unresectable and/or metastatic) solid tumors, were recruited into a single arm.
Pre-assignment Details: Per protocol, response/progression or adverse events during the second pembrolizumab course were not counted towards efficacy outcome measures or safety outcome measures respectively.
  Per protocol, analyses of disease type cohort was planned and conducted for efficacy outcome measures only.
Groups:
- Pembrolizumab 10 mg/kg: Participants received pembrolizumab 10 mg/kg intravenously (IV) over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. Qualified participants who completed the first course of pembrolizumab treatment but progressed after discontinuation were eligible for a second course of pembrolizumab at 10 mg/kg IV Q2W for up to ~1 additional year, at the Investigator's discretion. Per protocol participants were presented by treatment received in the single arm study.
Period: Overall Study
Arm/Group | Pembrolizumab 10 mg/kg
Started | 477
Treated During First Course | 475
Treated During Second Course | 11
Completed | 0
Not Completed | 477
Not completed — Sponsor Decision | 31
Not completed — Withdrawal by Subject | 43
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 10
Not completed — Death | 391

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all allocated participants who received at least one dose of study drug. Per protocol, Baseline Characteristics were summarized by treatment dose.
Groups:
- Pembrolizumab (MK-3475) 10 mg/kg: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. Qualified participants who completed the first course of pembrolizumab treatment but progressed after discontinuation were eligible for a second course of pembrolizumab at 10 mg/kg IV Q2W for up to ~1 additional year, at the Investigator's discretion. Per protocol participants were presented by treatment received in the single arm study.
Arm/Group | Pembrolizumab (MK-3475) 10 mg/kg
Number analyzed (Participants) | 475
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281
  Male | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 380
  Unknown or Not Reported | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 99
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 280
  More than one race | 2
  Unknown or Not Reported | 73

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) was defined as the percentage of participants who experienced a complete response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by the investigator.
Time Frame: Up to approximately 86 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, had a baseline scan with measurable disease per modified RECIST 1.1 and had the intended indication. Per protocol, participants were analyzed according to disease type.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort A1: Colon or Rectal Adenocarcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with colon or rectal adenocarcinoma.
- Cohort A2: Anal Canal Squamous Cell Carcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with anal canal squamous cell carcinoma.
- Cohort A3: Pancreas Adenocarcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with pancreas adenocarcinoma.
- Cohort A4: Esophageal Squamous Cell Carcinoma or Adenocarcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with esophageal squamous cell carcinoma or adenocarcinoma (including gastroesophageal (GE) junction).
- Cohort A5: Biliary Tract Adenocarcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with biliary tract adenocarcinoma (gallbladder and biliary tree, but excluding ampulla of vater cancers).
- Cohort A6: Carcinoid Tumors: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with carcinoid tumors.
- Cohort A7: Neuroendocrine Carcinomas: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with neuroendocrine carcinomas (well or moderately differentiated pancreatic neuroendocrine tumor).
- Cohort B1: ER Positive HER2 Negative Breast Cancer: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with estrogen receptor (ER) positive human epidermal growth factor receptor (HER2) negative breast cancer.
- Cohort B2: Ovarian Epithelial, Fallopian Tube or Primary Peritoneal Carcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with ovarian epithelial, fallopian tube or primary peritoneal carcinoma.
- Cohort B3: Endometrial Carcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with endometrial carcinoma.
- Cohort B4: Cervical Squamous Cell Cancer: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with cervical squamous cell cancer.
- Cohort B5: Vulvar Squamous Cell Carcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with vulvar squamous cell carcinoma.
- Cohort C1: Small Cell Lung Cancer: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with small cell lung cancer.
- Cohort C2: Mesothelioma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with mesothelioma (malignant pleural mesothelioma).
- Cohort D1: Thyroid Cancer: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with thyroid cancer (papillary or follicular subtype).
- Cohort D2: Salivary Gland Carcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with salivary gland carcinoma.
- Cohort D3: Nasopharyngeal Carcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with nasopharyngeal carcinoma.
- Cohort E1: Glioblastoma Multiforme: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with glioblastoma multiforme.
- Cohort E2: Leiomyosarcoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with leiomyosarcoma.
- Cohort E3: Prostate Adenocarcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with prostate adenocarcinoma.
Arm/Group | Cohort A1: Colon or Rectal Adenocarcinoma | Cohort A2: Anal Canal Squamous Cell Carcinoma | Cohort A3: Pancreas Adenocarcinoma | Cohort A4: Esophageal Squamous Cell Carcinoma or Adenocarcinoma | Cohort A5: Biliary Tract Adenocarcinoma | Cohort A6: Carcinoid Tumors | Cohort A7: Neuroendocrine Carcinomas | Cohort B1: ER Positive HER2 Negative Breast Cancer | Cohort B2: Ovarian Epithelial, Fallopian Tube or Primary Peritoneal Carcinoma | Cohort B3: Endometrial Carcinoma | Cohort B4: Cervical Squamous Cell Cancer | Cohort B5: Vulvar Squamous Cell Carcinoma | Cohort C1: Small Cell Lung Cancer | Cohort C2: Mesothelioma | Cohort D1: Thyroid Cancer | Cohort D2: Salivary Gland Carcinoma | Cohort D3: Nasopharyngeal Carcinoma | Cohort E1: Glioblastoma Multiforme | Cohort E2: Leiomyosarcoma | Cohort E3: Prostate Adenocarcinoma
Number analyzed (Participants) | 23 | 25 | 24 | 23 | 23 | 25 | 16 | 25 | 26 | 23 | 24 | 18 | 23 | 25 | 22 | 26 | 27 | 25 | 24 | 23
Percentage of Participants | 4.3 [0.1 to 21.9] | 20.0 [6.8 to 40.7] | 0.0 [0.0 to 14.2] | 30.4 [13.2 to 52.9] | 17.4 [5.0 to 38.8] | 16.0 [4.5 to 36.1] | 6.3 [0.2 to 30.2] | 12.0 [2.5 to 31.2] | 11.5 [2.4 to 30.2] | 13.0 [2.8 to 33.6] | 16.7 [4.7 to 37.4] | 5.6 [0.1 to 27.3] | 34.8 [16.4 to 57.3] | 20.0 [6.8 to 40.7] | 13.6 [2.9 to 34.9] | 11.5 [2.4 to 30.2] | 25.9 [11.1 to 46.3] | 8.0 [1.0 to 26.0] | 4.2 [0.1 to 21.1] | 13.0 [2.8 to 33.6]

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants with at least one AE was assessed.
Time Frame: Up to approximately 28 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab (MK-3475) 10 mg/kg: Participants received pembrolizumab 10 mg/kg intravenously (IV) over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. Per protocol participants were presented by treatment received in the single arm study.
Arm/Group | Pembrolizumab (MK-3475) 10 mg/kg
Number analyzed (Participants) | 475
Participants | 456

3. Secondary Outcome: Number of Participants Who Discontinued From Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued treatment due to an AE was assessed.
Time Frame: Up to approximately 25 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab (MK-3475) 10 mg/kg
Number analyzed (Participants) | 475
Participants | 30

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of allocation to the date of the first documentation of disease progression, as determined by investigator per modified RECIST 1.1 or death due to any cause (whichever occurred first). Disease progression was defined as at least 20 percent (%) increase (including an absolute increase of at least 5 millimeter [mm]) in the sum of diameter of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. PFS was estimated and analyzed using Kaplan-Meier method.
Time Frame: Up to approximately 86 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort B1: ER Positive HER2 Negative Breast Cancer: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with ER positive HER2 negative breast cancer.
Arm/Group | Cohort A1: Colon or Rectal Adenocarcinoma | Cohort A2: Anal Canal Squamous Cell Carcinoma | Cohort A3: Pancreas Adenocarcinoma | Cohort A4: Esophageal Squamous Cell Carcinoma or Adenocarcinoma | Cohort A5: Biliary Tract Adenocarcinoma | Cohort A6: Carcinoid Tumors | Cohort A7: Neuroendocrine Carcinomas | Cohort B1: ER Positive HER2 Negative Breast Cancer | Cohort B2: Ovarian Epithelial, Fallopian Tube or Primary Peritoneal Carcinoma | Cohort B3: Endometrial Carcinoma | Cohort B4: Cervical Squamous Cell Cancer | Cohort B5: Vulvar Squamous Cell Carcinoma | Cohort C1: Small Cell Lung Cancer | Cohort C2: Mesothelioma | Cohort D1: Thyroid Cancer | Cohort D2: Salivary Gland Carcinoma | Cohort D3: Nasopharyngeal Carcinoma | Cohort E1: Glioblastoma Multiforme | Cohort E2: Leiomyosarcoma | Cohort E3: Prostate Adenocarcinoma
Number analyzed (Participants) | 23 | 25 | 24 | 23 | 23 | 25 | 16 | 25 | 26 | 23 | 24 | 18 | 23 | 25 | 22 | 26 | 27 | 25 | 24 | 23
Months | 1.7 [1.4 to 1.8] | 3.1 [1.6 to 6.2] | 1.7 [1.5 to 1.8] | 1.8 [1.7 to 2.9] | 1.8 [1.4 to 2.1] | 5.5 [3.5 to 10.7] | 4.5 [3.5 to 13.9] | 1.8 [1.4 to 3.6] | 1.9 [1.8 to 3.5] | 1.8 [1.6 to 2.7] | 1.8 [1.6 to 3.2] | 2.5 [1.4 to 3.7] | 1.8 [1.7 to 5.8] | 5.5 [3.5 to 8.2] | 8.2 [2.2 to 14.4] | 3.6 [1.8 to 5.1] | 6.4 [3.5 to 13.4] | 2.8 [1.9 to 8.1] | 2.0 [1.7 to 5.3] | 3.5 [1.7 to 6.5]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of allocation to the date of death due to any cause. Participants who were lost to follow-up and those who were alive at the end of the trial were censored at the date of last assessment.
Time Frame: Up to approximately 86 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort B1: HR Positive HER2 Negative Breast Cancer: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled with ER positive HER2 negative breast cancer.
Arm/Group | Cohort A1: Colon or Rectal Adenocarcinoma | Cohort A2: Anal Canal Squamous Cell Carcinoma | Cohort A3: Pancreas Adenocarcinoma | Cohort A4: Esophageal Squamous Cell Carcinoma or Adenocarcinoma | Cohort A5: Biliary Tract Adenocarcinoma | Cohort A6: Carcinoid Tumors | Cohort A7: Neuroendocrine Carcinomas | Cohort B1: HR Positive HER2 Negative Breast Cancer | Cohort B2: Ovarian Epithelial, Fallopian Tube or Primary Peritoneal Carcinoma | Cohort B3: Endometrial Carcinoma | Cohort B4: Cervical Squamous Cell Cancer | Cohort B5: Vulvar Squamous Cell Carcinoma | Cohort C1: Small Cell Lung Cancer | Cohort C2: Mesothelioma | Cohort D1: Thyroid Cancer | Cohort D2: Salivary Gland Carcinoma | Cohort D3: Nasopharyngeal Carcinoma | Cohort E1: Glioblastoma Multiforme | Cohort E2: Leiomyosarcoma | Cohort E3: Prostate Adenocarcinoma
Number analyzed (Participants) | 23 | 25 | 25 | 23 | 24 | 25 | 16 | 25 | 26 | 24 | 24 | 18 | 23 | 25 | 22 | 26 | 27 | 26 | 24 | 23
Months | 5.3 [2.2 to 10.9] | 8.3 [5.8 to 16.2] | 3.9 [2.8 to 5.5] | 7.1 [4.3 to 17.7] | 5.7 [3.1 to 9.8] | 16.2 [7.6 to 22.4] | 37.8 [20.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 8.0 [6.5 to 10.3] | 13.1 [7.3 to 18.8] | 13.6 [2.2 to 25.2] | 10.8 [3.8 to 15.4] | 3.7 [3.1 to 7.7] | 9.3 [4.1 to 10.6] | 18.0 [10.3 to 24.4] | 39.7 [29.7 to 65.0] | 12.3 [6.0 to 30.1] | 16.5 [10.1 to 31.9] | 13.1 [8.0 to 26.6] | 12.0 [7.7 to 18.3] | 7.9 [6.5 to 15.3]

6. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per modified RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per modified RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. DOR assessments were based on investigator with confirmation. The DOR according to modified RECIST 1.1 for all participants who experienced a confirmed CR or PR was reported. Per protocol, participants were analyzed according to disease type.
Time Frame: Up to approximately 86 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, had a baseline scan with measurable disease per modified RECIST 1.1, had the intended indication, and experienced a response. Per protocol-specified definition, DOR could not be analyzed in arms which did not have a confirmed response of CR or PR.
Measure: Median (Full Range); unit: Months
Groups:
- Cohort B3: Endometrial Carcinoma: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled endometrial carcinoma.
- Cohort B4: Cervical Squamous Cell Cancer: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years. This cohort represents all participants who enrolled cervical squamous cell cancer.
Arm/Group | Cohort A1: Colon or Rectal Adenocarcinoma | Cohort A2: Anal Canal Squamous Cell Carcinoma | Cohort A3: Pancreas Adenocarcinoma | Cohort A4: Esophageal Squamous Cell Carcinoma or Adenocarcinoma | Cohort A5: Biliary Tract Adenocarcinoma | Cohort A6: Carcinoid Tumors | Cohort A7: Neuroendocrine Carcinomas | Cohort B1: ER Positive HER2 Negative Breast Cancer | Cohort B2: Ovarian Epithelial, Fallopian Tube or Primary Peritoneal Carcinoma | Cohort B3: Endometrial Carcinoma | Cohort B4: Cervical Squamous Cell Cancer | Cohort B5: Vulvar Squamous Cell Carcinoma | Cohort C1: Small Cell Lung Cancer | Cohort C2: Mesothelioma | Cohort D1: Thyroid Cancer | Cohort D2: Salivary Gland Carcinoma | Cohort D3: Nasopharyngeal Carcinoma | Cohort E1: Glioblastoma Multiforme | Cohort E2: Leiomyosarcoma | Cohort E3: Prostate Adenocarcinoma
Number analyzed (Participants) | 1 | 5 | 0 | 7 | 4 | 4 | 1 | 3 | 3 | 3 | 4 | 1 | 8 | 5 | 3 | 3 | 7 | 2 | 1 | 3
Months | NA [NA to NA] — NA = Median, upper limit, lower limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 28.9 [3.8 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. |  | 14.5 [5.6 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [6.0 to NA] — NA = Median, upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 10.1 [6.9 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 25.1 [25.1 to 25.1] | 12.0 [7.4 to 15.9] | 37.0 [34.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 68.5 [17.5 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 5.4 [4.1 to 7.5] | 3.9 [3.9 to 3.9] | NA [NA to NA] — NA = Median, upper limit, lower limit not reached at time of data cut-off due to insufficient number of responding participants with relapse. | 12.0 [3.7 to 44.4] | 8.4 [4.6 to 20.3] | 3.9 [3.5 to 20.6] | 15.0 [4.8 to 34.0] | 15.6 [8.3 to 22.8] | 12.4 [12.4 to 12.4] | 14.2 [13.5 to 31.4]

ADVERSE EVENTS:
Time Frame: Up to ~28 months for first course and up to ~49 months for second course. All-cause mortality (ACM): Up to ~86 months for first and second course.
Description: ACM includes all randomized participants. Safety includes all participants receiving ≥1 dose of study treatment. Per protocol, AEs were collected and reported by treatment intervention irrespective of indication. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs. Participants receiving a second course of pembrolizumab per protocol were monitored for ACM and safety separately.
Groups:
- First Course Pembrolizumab 10 mg/kg: Participants received pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years.
- Second Course Pembrolizumab 10 mg/kg: Qualified participants who completed the first course of pembrolizumab 10 mg/kg IV over 30 minutes once every 2 weeks (Q2W) for up to ~2 years, but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 10 mg/kg IV Q2W for up to ~1 year.
Arm/Group | First Course Pembrolizumab 10 mg/kg | Second Course Pembrolizumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 426/477 | 6/11
Serious Adverse Events (participants affected / at risk) | 160/475 | 3/11
Other Adverse Events (participants affected / at risk) | 429/475 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Course Pembrolizumab 10 mg/kg (N=475) | Second Course Pembrolizumab 10 mg/kg (N=11)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 7 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 4 (4) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 8 (11) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (4) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (2) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Ureteric dilatation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Noninfective bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | First Course Pembrolizumab 10 mg/kg (N=475) | Second Course Pembrolizumab 10 mg/kg (N=11)
Anaemia (Blood and lymphatic system disorders) | 87 (101) | 0 (0)
Hypothyroidism (Endocrine disorders) | 38 (39) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 54 (59) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 28 (31) | 1 (1)
Constipation (Gastrointestinal disorders) | 93 (105) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 102 (177) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 29 (30) | 1 (1)
Nausea (Gastrointestinal disorders) | 124 (149) | 0 (0)
Vomiting (Gastrointestinal disorders) | 75 (99) | 1 (1)
Asthenia (General disorders) | 59 (68) | 1 (1)
Fatigue (General disorders) | 165 (176) | 0 (0)
Oedema peripheral (General disorders) | 43 (47) | 1 (1)
Pyrexia (General disorders) | 74 (97) | 0 (0)
Alanine aminotransferase increased (Investigations) | 31 (39) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 37 (45) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 40 (41) | 0 (0)
Weight decreased (Investigations) | 35 (36) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 102 (106) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 35 (37) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 31 (33) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 37 (46) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 34 (36) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 77 (101) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 56 (64) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 38 (49) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 (34) | 0 (0)
Dizziness (Nervous system disorders) | 42 (54) | 0 (0)
Headache (Nervous system disorders) | 63 (73) | 1 (1)
Depression (Psychiatric disorders) | 25 (26) | 0 (0)
Insomnia (Psychiatric disorders) | 44 (45) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 69 (89) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 60 (67) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 24 (25) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 69 (88) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 56 (71) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 25 (28) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 8 (9) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 4 (7) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (13) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 18 (18) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (3) | 1 (1)
Hematuria (Renal and urinary disorders) | 10 (19) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3/11 (5) | 1 (1)
Hypotension (Vascular disorders) | 20 (21) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Conjunctivitis (Infections and infestations) | 7 (7) | 2 (2)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 7 (7) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 21 (27) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 7 (7) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 14 (19) | 2 (2)
Chest pain (General disorders) | 20 (23) | 1 (1)
Influenza like illness (General disorders) | 11 (16) | 2 (3)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 5 (5) | 1 (1)
Dry eye (Eye disorders) | 11 (11) | 2 (2)
Uveitis (Eye disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT02054806/Prot_SAP_000.pdf